CLINICAL TRIAL: NCT03048370
Title: Reactivity of the Vestibular System to Caloric Vestibular Stimulation in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Philip Gerretsen, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 042-2016
Record Dates: First submitted 2016-12-14; First posted 2017-02-09 (Estimated); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Schizophrenia; Healthy
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: Each participant will successively receive 6 vestibular stimulation conditions. Side of stimulation will be randomized.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will be blinded to the order of experimental conditions, as well as the person conducting specific ratings assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Left body temperature VS (Experimental): Left body temperature (37°C) vestibular stimulation
  Interventions: Procedure: Left body temperature VS
- Right body temperature VS (Experimental): Right body temperature (37°C) vestibular stimulation
  Interventions: Procedure: Right body temperature VS
- Left warm CVS (Experimental): Left warm (44°C) caloric vestibular stimulation
  Interventions: Procedure: Left warm CVS
- Right warm CVS (Experimental): Right warm (44°C) caloric vestibular stimulation
  Interventions: Procedure: Right warm CVS
- Left cold CVS (Experimental): Left cold (30°C) caloric vestibular stimulation
  Interventions: Procedure: Left cold CVS
- Right cold CVS (Experimental): Right cold (30°C) caloric vestibular stimulation
  Interventions: Procedure: Right cold CVS

INTERVENTIONS:
Procedure: Left body temperature VS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Left body temperature VS
Procedure: Right body temperature VS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Right body temperature VS
Procedure: Left warm CVS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Left warm CVS
Procedure: Right warm CVS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Right warm CVS
Procedure: Left cold CVS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Left cold CVS
Procedure: Right cold CVS — Caloric vestibular stimulation (CVS), which involves the irrigation of cold or warm water into the external ear canal, induces a temperature gradient across the semicircular canals of the vestibular apparatus stimulating the vestibular nerve. It is commonly used in both otolaryngology to assess vestibular function and neurology to test brain stem function
  Arms: Right cold CVS

SUMMARY:
This study aims to determine if individuals with schizophrenia have greater reactivity to vestibular stimulation than healthy controls. The physiological response of vestibular stimulation will be assessed with electronystagmography, which provides a measure of the intensity of the nystagmus via PSPV. Positive results would suggest greater vestibular system reactivity to vestibular stimulation may be a biomarker of schizophrenia. Pathophysiologically, increased vestibular reactivity to vestibular stimulation may reflect abnormal vestibular function or impaired central suppression of the vestibular ocular reflex.

DETAILED DESCRIPTION:
In schizophrenia, there is no conclusive link between psychopathology and vestibular dysfunction and we are not aware of any data that exists on the range of responses to caloric vestibular stimulation (CVS) in persons with schizophrenia. Initial data from another CVS study from our group suggests individuals with schizophrenia have greater reactivity to body temperature (37°C) CVS, as measured by the peak slow phase velocity of the resulting nystagmus (PSPV), than would be expected from individuals without schizophrenia versus healthy participants. Intriguingly, CVS at 37°C should not theoretically produce a significant vestibulocular reflex response due to the stimulus' approximation to body temperature. Hence, the primary aim of this study is to determine if individuals with schizophrenia will have greater vestibular reactivity, as measured by nystagmus PSPV, to CVS in comparison with healthy participants. The secondary aim is to assess illness awareness pre and post CVS administration in attempts to replicate our previous observation. A total of 20 patients with schizophrenia and 20 healthy control participants will be recruited. All participants will receive three conditions bilaterally: (1) body temperature (37°C) vestibular stimulation; (2) warm CVS (44°C), and (3) cold CVS (30°C).

ELIGIBILITY:
Inclusion Criteria for Schizophrenia group:

1. Male or female inpatients or outpatients age ≥18
2. Having a DSM-5 diagnosis of schizophrenia or schizoaffective disorder
3. Voluntary and capable of consenting to participation in the research study
4. Fluent in English

Inclusion Criteria for Healthy Controls group:

1. Male or female and age ≥18
2. Voluntary and capable of consenting to participation in the research study
3. Fluent in English
4. Absence of history of psychiatric illness using the Mini-International Neuropsychiatric Interview (MINI)

Exclusion Criteria for all participants:

1. Serious unstable medical illness or any concomitant major medical or neurological illness
2. Acute suicidal and/or homicidal ideation
3. Formal thought disorder rating of over 2 on the Scale for Assessment of Positive Symptoms (SAPS) [patients only]
4. DSM-IV substance dependence (except caffeine and nicotine) within one month prior to entering the study
5. Pregnant women
6. Positive urine drug screen
7. History of external or middle ear pathology
8. History or signs of middle ear surgery (e.g. Tympanoplasty, mastoidectomy)
9. Signs of active ear disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Nystagmus response (peak slow phase velocity) | Between 30 and 60 sec after each CVS condition
  Nystagmus response will be measured at between thirty and 60 seconds post irrigations, looking for the highest velocities.

SECONDARY OUTCOMES:
Illness awareness | Before CVS session and10 min after CVS session
  Changes in illness awareness will be assessed using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Gerretsen, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.net/research